CLINICAL TRIAL: NCT02139111
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Parallel-Arm, Multi-Center Study Measuring the Efficacy and Safety of PRC-063 in Adolescent ADHD Patients
Brief Title: PRC-063 in Adolescent ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rhodes Pharmaceuticals, L.P. (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 063-009
Record Dates: First submitted 2014-05-12; First posted 2014-05-15 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo Arm
  Interventions: Drug: Placebo
- PRC-063 25 mg and Placebo (Active Comparator): PRC-063 25 mg and placebo capsule by mouth once daily
  Interventions: Drug: Placebo; Drug: PRC-063 25 mg
- PRC-063 45 mg and Placebo (Active Comparator): PRC-063 45 mg and placebo capsule by mouth once daily
  Interventions: Drug: Placebo; Drug: PRC-063 45 mg
- PRC-063 70 mg and Placebo (Active Comparator): PRC-063 70 mg and placebo capsule by mouth once daily
  Interventions: Drug: Placebo; Drug: PRC-063 70 mg
- PRC-063 85 mg and Placebo (Active Comparator): PRC-063 85 mg and placebo capsule by mouth once daily
  Interventions: Drug: Placebo; Drug: PRC-063 85 mg

INTERVENTIONS:
Drug: Placebo — Oral placebo capsule
  Other Names: Placebo capsule
Drug: PRC-063 25 mg — Oral 25 mg capsule - active
  Other Names: 25 mg capsule
  Arms: PRC-063 25 mg and Placebo
Drug: PRC-063 45 mg — Oral 45 mg capsule - active
  Other Names: 45 mg capsule
  Arms: PRC-063 45 mg and Placebo
Drug: PRC-063 70 mg — Oral 70 mg capsule - active
  Other Names: 70 mg capsule
  Arms: PRC-063 70 mg and Placebo
Drug: PRC-063 85 mg — Oral 85 mg capsule - active
  Other Names: 85 mg capsule
  Arms: PRC-063 85 mg and Placebo

SUMMARY:
The purpose of this randomized, placebo-controlled, double-blind, parallel group study is to evaluate the clinical efficacy and safety of PRC-063 in adolescents with ADHD.

DETAILED DESCRIPTION:
This study is a randomized, phase III, multicenter, placebo-controlled, parallel-group, forced-dose titration in which adolescent subjects (12 to 17 years of age inclusive) with ADHD will be randomized to PRC-063 (25, 45, 70 or 85 mg) or placebo for four weeks of double-blind evaluation of safety and efficacy. The study will have four phases: (1) screening and 1-week washout; (2)baseline and double-blind, forced-dose titration over a 2-week period; (3) double-blind evaluation over a 2-week period; and (4) a 14-day safety follow-up. Subjects will be required to visit the site 6 times over a 5 week period.

Screening and Washout: Subjects will be screened to establish eligibility for study participation. Subjects who meet eligibility requirements will undergo ADHD medication washout, if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Must be male or non-pregnant female at least 12 years of age and less than 18 years of age.
* Must have an ADHD diagnosis, in attentive, hyperactive/impulsive or combined, as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) based on clinician assessment using multiple informants and a structured interview.
* Must be unsatisfied with his or her current pharmacological therapy for treatment of ADHD or not currently receiving pharmacological therapy for ADHD. Inclusion of subjects naïve to pharmacological therapy for ADHD is permitted.
* Female subjects must be one of the following: a. surgically sterile prior to screening; b. if of childbearing potential, abstinent or willing to use a reliable method of contraception, such as oral contraceptive, two barrier methods, a barrier method plus a spermicidal agent.
* Female subjects of Child-Bearing Potential (FOCP) must be a negative serum β-hCG pregnancy test at screening.
* Must have a minimum level of intellectual functioning, as determined by an Intelligence Quotient (IQ) score of 80 or above based on the WASI or the KBIT.
* Mentally and physically competent to sign an informed assent document, in the case of the subject, and an informed consent document, in the case of the parent/guardian, indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Able and willing to comply with the study procedures for the entire length of the study, including a successful swallow test of an empty 85 mg capsule.
* Total score of 24 or greater on the clinician-rated ADHA-5-RS, as assessed at Visit 2

Exclusion Criteria:

* Having an allergy to methylphenidate or amphetamines or a history of serious adverse reactions to methylphenidate.
* Known to be non-responsive to methylphenidate treatment. Non-response is defined as methylphenidate use at various doses for a phase of at least four weeks at each dose with little or no clinical benefit.
* Being diagnosed with or having a history of strokes, epilepsy, migraine headaches (greater than 1 instance every two months), glaucoma, thyrotoxicosis, tachyarrhythmias or severe angina pectoris or have serious or unstable medical illness. Subjects with controlled or stable asthma or diabetes will be permitted.
* Elevated blood pressure, defined as any values above 89 diastolic or 139 systolic, as assessed at Visit 1.
* Clinically significant ECG abnormalities, as assessed at Visit 1.
* Clinically significant laboratory abnormalities, as assessed at Visit 1.
* Currently receiving guanethidine, pressor agents, MAO inhibitors, coumarin anticoagulants, anticonvulsants (e.g., phenobarbital, phenytoin, primidone), phenylbutazone, tricyclic antidepressants (e.g., imipramine, desipramine), selective serotonin reuptake inhibitors (SSRIs) or herbal remedies (unless on a stable dose for 4 weeks).
* Subject has known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary heart disease, transient ischemic attack or stroke or other serious cardiac problems that may place the subject at increased vulnerability to the sympathomimetic effects of a stimulant drug.
* Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
* Subjects who are currently considered a suicide risk by the investigator.
* Having a primary diagnosis of schizophrenia, schizoaffective disorder, primary affective disorder, schizotypal personality, major depression, bipolar disorder, generalized anxiety, borderline personality disorder, antisocial personality or another unstable psychiatric condition requiring treatment, as assessed by the structured interview conducted at Visit 1.
* Having a history or suspected physiological dependence (excluding nicotine) on narcotic analgesics or other psychoactive drugs (including barbiturates, opiates, cocaine, cannabinoids, amphetamines and benzodiazepines).
* Excessive consumption of alcohol (consumes alcohol in quantities greater than 15 drinks per week; 1 drink is defined as 360 mL/12 oz. of beer, 120 mL/4 oz. of wine, or 30 mL/1 oz. of hard liquor), or history (within previous 6 months) of alcohol abuse.
* Currently (or within 30 days before the planned start of treatment) receiving an investigational drug or using an experimental medical device.
* Homeless.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Clinician-administered ADHD-5-Rating Scale | Baseline week 2, weeks 3-6

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Reiz, Study Director — Purdue Pharma LP
Locations (43):
- United States (31):
  - UCLA, Los Angeles, California
  - Synergy Clinical Research, National City, California
  - Newport Beach Clinical Research Associates, Inc., Newport Beach, California
  - Orange County Neuro Phychiatry Research Centre, Orange, California
  - Florida Clinical Research Center, Bradenton, Florida
  - Sarkis Clinical Research, Gainesville, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - CNS Healthcare Jacksonville, Jacksonville, Florida
  - Florida Clinical Research Center, Maitlin, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Advanced Clinical Research, Boise, Idaho
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Center for Psychiatry and Behavioral Medicine Inc., Las Vegas, Nevada
  - Duke University Medical Center, Durham, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - FutureSearch Clinical Trials, L.P., Austin, Texas
  - FutureSearch Trials of Dallas, L.P., Dallas, Texas
  - Bayou City Research Ltd, Houston, Texas
  - Red Oak Psychiatry Associates, Houston, Texas
  - Houston Clinical Trials, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Ericksen Research, Clinton, Utah
  - Physiciatric and Behavioral Solutions, Salt Lake City, Utah
  - NeuroScience, Herndon, Virginia
  - Northwest Clinical Research Center, Friday Harbor, Washington
  - Eastside Therapeutic Resource, Kirkland, Washington
- Canada (12):
  - Mathison Centre for Mental Health Research and Education, Calgary, Alberta
  - University of Calgary, Calgary, Alberta
  - Chokka Center for Integrative Health, Edmonton, Alberta
  - Dr. Margaret Weiss, Vancouver, British Columbia
  - Atlantic ADHD Centre, Dartmouth, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Doctors Jackiewicz Professional Medical Corporation, Niagra Falls, Ontario
  - Dr. Judy van Stralen, Ottawa, Ontario
  - Stress, Trauma, Anxiety, Rehabilitation and Treatment (START) in the Mood and Anxiety Disorders Clinic, Toronto, Ontario
  - The Kids Clinic, Whitby, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Royal University Hospital Saskatoon, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Storebo OJ, Storm MRO, Pereira Ribeiro J, Skoog M, Groth C, Callesen HE, Schaug JP, Darling P, Huus CL, Zwi M, Kirubakaran R, Simonsen E, Gluud C. Methylphenidate for children and adolescents with attention deficit hyperactivity disorder (ADHD). Cochrane Database Syst Rev. 2025 Dec 4;12(12):CD009885. doi: 10.1002/14651858.CD009885.pub4. PMID 41342306
- [Derived] Storebo OJ, Storm MRO, Pereira Ribeiro J, Skoog M, Groth C, Callesen HE, Schaug JP, Darling Rasmussen P, Huus CL, Zwi M, Kirubakaran R, Simonsen E, Gluud C. Methylphenidate for children and adolescents with attention deficit hyperactivity disorder (ADHD). Cochrane Database Syst Rev. 2023 Mar 27;3(3):CD009885. doi: 10.1002/14651858.CD009885.pub3. PMID 36971690
- [Derived] Weiss MD, Surman C, Khullar A, Owens J, He E, Cataldo M, Donnelly G. Effect of a Multilayer, Extended-Release Methylphenidate Formulation (PRC-063) on Sleep in Adolescents with Attention-Deficit/Hyperactivity Disorder: A Randomized, Double-Blind, Fixed-Dose, Placebo-Controlled Trial Followed by a 6-Month Open-Label Follow-Up. J Child Adolesc Psychopharmacol. 2021 Nov;31(9):623-630. doi: 10.1089/cap.2021.0087. Epub 2021 Oct 28. PMID 34714112
- [Derived] Weiss MD, Cutler AJ, Kollins SH, Donnelly GAE. Efficacy and Safety of a Long-Acting Multilayer-Release Methylphenidate Formulation (PRC-063) in the Treatment of Adolescent Attention-Deficit/Hyperactivity Disorder: A Randomized, Double-Blind Clinical Trial with a 6-Month Open-Label Extension. J Child Adolesc Psychopharmacol. 2021 Nov;31(9):610-622. doi: 10.1089/cap.2021.0034. Epub 2021 Oct 8. PMID 34637343